CLINICAL TRIAL: NCT02100241
Title: Effectiveness Analysis of Active Stretching Versus Active Stretching With Low Frequency Currents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodríguez, Francisco Piqueras, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPR2012
Record Dates: First submitted 2013-07-19; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Muscular Diseases
Keywords: Young adult; Muscle Stretching Exercises; Range of Motion, Articular
MeSH Terms: conditions — Muscular Diseases | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active stretching with currents (Experimental): Active stretching performed while currents are applied on hamstring muscles.
  Interventions: Procedure: Active stretching
- Active stretching (Experimental): Active stretching are performed.
  Interventions: Procedure: Active stretching
- Control group (No Intervention): Routine clinical practice

INTERVENTIONS:
Procedure: Active stretching — The participants performed three specific exercises of static active stretching of the hamstring muscles, maintaining the maximum tightness that was tolerable without pain for 15 seconds. Each exercise were performed twice, with a total of six repetitions.
  Arms: Active stretching; Active stretching with currents

SUMMARY:
The purpose of this study is to determine whether active stretching with low frequency currents are more effective than active stretching in the treatment of hamstring shortness syndrome in children.

DETAILED DESCRIPTION:
In 2012 we studied 51 young footballers with Short Hamstring Syndrome in Spain. Three groups were formed:

1. Stretching+Transcutaneous Electrical Nervous Stimulation (TENS);
2. Active stretching;
3. Conventional stretching.

Parameters: straight leg raise test (SLR), popliteal angle with the passive knee extension test (PKE) and the toe-touch test (TT).

The inter-group means were compared and clinically relevant parameters calculated [relative risk (RR), absolute risk reduction (ARR), relative risk reduction (RRR) and number needed to treat (NNT)].

ELIGIBILITY:
Inclusion Criteria:

* children between 10 to 16.
* children federated belonging to Football School of Jumilla.
* children whose result in the assessment of range of motion is less than 70º in the Straight Leg Raising Test.
* not afraid to present the application of electrotherapy.
* not have low back pain in last three months.
* not to be injured

Exclusion Criteria:

* children who have acute muscle injury or ligamentous.
* children with recent fractures or unconsolidated.
* children with ligamentous laxity.
* functional shortening suffering children

Ages: 10 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Range of motion | a week

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Piqueras, PT, Principal Investigator
Locations (1):
- Universidad Miguel Hernandez de Elche, Sant Joan d'Alacant, Alicante, Spain